CLINICAL TRIAL: NCT06588673
Title: Art Therapy in Progressive Supranuclear Palsy: Studying the Effect on Quality of Care
Brief Title: Art Therapy in Progressive Supranuclear Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: CurePSP Foundation (Unknown)
Responsible Party: Principal Investigator, Amy E Brown, Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 240791
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art Therapy (Other): psp patients enrolled into study.
  Interventions: Other: Art Thrapy

INTERVENTIONS:
Other: Art Thrapy — Art therapy at Art Therapy Studio, a well-established recommended art therapy leader since 1967 with extensive experience in virtual therapy for patients with medical needs. Cheryl Pete, MA ATR-BC, a board-certified art therapist and the Clinical Director will complete the art therapy sessions. The art therapy will be a 1-hour sessions, once a week for a total of 8 weeks (or 8 sessions). Cheryl Pete's role will solely involve providing a service. Chery will complete the Art Therapy according to her standard practices. Cheryl's Art Therapy will not be altered in any way as a part of this research study. Cheryl will not collect any research data. As research participants are referred to Cheryl for the Art Therapy, the research participant's name and contact information will be shared.

SUMMARY:
Our aim is to study the effect of art therapy for people with PSP, with a focus on alleviating the symptoms associated with PSP, enhancing the overall quality of life for patients, and reducing caregiver stress. Overall, through our collaborative efforts on this study, we hope to unlock the benefits of art therapy for this vulnerable patient population, ultimately improving their overall well-being and enhancing their quality of life.

DETAILED DESCRIPTION:
Progressive Supranuclear Palsy (PSP) is typically manifested by a multitude of distressing symptoms, including bradyphrenia and bradykinesia, speech dyspraxia, visual problems, and postural instability with high risk of falls. These symptoms not only inflict physical hardships on patients but also have profound emotional and psychological implications. Thus, a decline in self-esteem, a reduction in the quality of life, and heightened stress for caregivers is remarkable. In recent years, art therapy has garnered attention as a potentially effective intervention for individuals grappling with neurodegenerative disorders. Art therapy encompasses a wide array of activities that promote cognitive and motor skills, including shape recognition, motion perception, sensory-motor integration, abstraction, and eye-hand coordination. As a result, it holds promise as a therapeutic tool for addressing the intricate challenges faced by PSP people. Although art therapy has demonstrated positive outcomes in enhancing visual cognitive skills, refining visual exploration strategies, and bolstering general motor function in Parkinson's disease, its potential in the context of PSP remains largely unexplored. Given the unique symptomatology and emotional toll of PSP, patients suffering from this condition stand to benefit significantly from the healing and therapeutic effects of art therapy. In light of these considerations, our proposal aims to bridge this knowledge gap by implementing and rigorously studying the impact of art therapy on PSP patients. Our aim is to investigate the effect of art therapy for people with PSP, with a focus on alleviating the symptoms associated with PSP, enhancing the overall quality of life for patients, and reducing caregiver stress. Overall, through our collaborative efforts on this study, we hope to unlock the benefits of art therapy for this vulnerable patient population, ultimately improving their overall well-being and enhancing their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of progressive supranuclear palsy
* Have the cognitive ability to provide informed consent

Exclusion Criteria:

* Primary neurological diagnosis other than progressive supranuclear palsy
* Cognition too impaired to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
PSP-QoL (Progressive Supranuclear Palsy Qualify of Life Scale) | 8-10 weeks
  Self-reported quality of life rating scale comprising of 28 items in six categories: daily activities (by history), behavior, bulbar, ocular motor, limb motor and gait/midline. Scores range from 0 to 100, each item graded 0-2 (six items) or 0-4 (22 items). The lower the total score the better the quality of life.

SECONDARY OUTCOMES:
PHQ-9 (Patient Health Questionnaire-9) | 8-10 weeks
  Self-reported depression rating scale comprising of 9 items. The lower the total score means that depression is absent or minimal.
NPI (Neuropsychiatric Inventory) | 8-10 weeks
  Scale that is completed by the caregiver. The scale is comprised of 12 items and will evaluate behavioral areas commonly affected in patients with dementia. The lower the total score means that behavior is intact
Zarit Caregiver Burden Scale | 8-10 weeks
  Scale that is completed by the caregiver. The scale is comprised of 22 items and will evaluate the caregiver's level of burden. The lower the total score means that the burden is absent.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
All data for the project will be coded. All coded IPD with be shared between Baylor and Vanderbilt will also be coded. Baylor University Neurology department is conducting their own PSP art therapy study in conjunction with VUMC. Each site will obtain their own local IRB approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 1 week of enrolling our first participant IPD will be shared. No expiration of this data.

REFERENCES:
- [Background] Cucca A, Acosta I, Berberian M, Lemen AC, Rizzo JR, Ghilardi MF, Quartarone A, Feigin AS, Di Rocco A, Biagioni MC. Visuospatial exploration and art therapy intervention in patients with Parkinson's disease: an exploratory therapeutic protocol. Complement Ther Med. 2018 Oct;40:70-76. doi: 10.1016/j.ctim.2018.07.011. Epub 2018 Jul 27. PMID 30219472
- [Background] Yu J, Rawtaer I, Goh LG, Kumar AP, Feng L, Kua EH, Mahendran R. The Art of Remediating Age-Related Cognitive Decline: Art Therapy Enhances Cognition and Increases Cortical Thickness in Mild Cognitive Impairment. J Int Neuropsychol Soc. 2021 Jan;27(1):79-88. doi: 10.1017/S1355617720000697. Epub 2020 Aug 7. PMID 32762792
- [Background] Cucca A, Di Rocco A, Acosta I, Beheshti M, Berberian M, Bertisch HC, Droby A, Ettinger T, Hudson TE, Inglese M, Jung YJ, Mania DF, Quartarone A, Rizzo JR, Sharma K, Feigin A, Biagioni MC, Ghilardi MF. Art therapy for Parkinson's disease. Parkinsonism Relat Disord. 2021 Mar;84:148-154. doi: 10.1016/j.parkreldis.2021.01.013. Epub 2021 Jan 23. PMID 33526323
- [Background] Perez Matos JA, Richard A, Spee BT, Pelowski M. Neurodegenerative diseases, art and creativity: therapeutic implications. Neurodegener Dis Manag. 2021 Jun;11(3):187-192. doi: 10.2217/nmt-2021-0012. Epub 2021 Jun 3. No abstract available. PMID 34078118